CLINICAL TRIAL: NCT04086511
Title: PANDA: A Cross-sectional Study to Measure Blood Amino Acid Levels in PKU Children on a Protein Substitute
Brief Title: PANDA: PKU Amino Acid Evaluation
Acronym: PANDA
Status: Completed | Type: Observational
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Other Study IDs: MBB18TA18444
Record Dates: First submitted 2019-09-10; First posted 2019-09-11 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2021-09

CONDITIONS: Phenylketonuria (PKU)
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with PKU
- Age- and sex-matched non-PKU comparison subjects

SUMMARY:
Phenylketonuria (PKU) is a rare inherited metabolic disorder, where subjects are born with a genetic deficiency in the phenylalanine hydroxylase enzyme (PAH), which leaves them unable to convert Phenylalanine (Phe) into Tyrosine (Tyr). PKU patients have specific dietary needs and must follow a restrictive diet in the aim of preventing toxic levels of the amino acid phenylalanine (Phe) accumulation.

DETAILED DESCRIPTION:
The exploratory study's main objective is to measure blood amino acid levels and to gain quantitative insights in children with PKU on a protein substitute with respect to evaluation of nutritional intake.

ELIGIBILITY:
Inclusion Criteria:

Both PKU and Non-PKU comparison subjects:

1. Age ≥ 2 and ≤ 12 years
2. Willing and able to provide informed consent by parents or legal representatives (and assent if required by local law/regulations)
3. One subject per family

   PKU subjects specific inclusion criteria:
4. PKU subjects identified by newborn screening and started low Phe diet before 1 month age
5. Usage of at least two Phe-free protein substitutes on a daily basis for at least 26 consecutive weeks up to Visit 1
6. Average Phe-level ≤360 µmol/L based on at least two blood Phe values from the past 12 months up to Visit 1

   Non-PKU comparison subjects specific inclusion criteria:
7. Same age (±3 years) and sex as an included PKU subject

Exclusion Criteria:

Both PKU and Non-PKU comparison subjects:

1. Current psychiatric disorders
2. Severe hepatic, thyroid or renal dysfunction
3. Acute illnesses like fever, flu, diarrhea, or vomiting (subjects should be symptom free for a week prior to V1)
4. Serious conditions (e.g. cancer, hydrocephalus, fatal heart disease)
5. Participation in any other clinical intervention studies involving test products concomitantly or within six weeks prior to entry into the study

   PKU specific exclusion criteria:
6. Use of BH4, or drugs that may interfere with main outcomes

   Non-PKU comparison subjects specific exclusion criteria:
7. PKU diagnosis or any other diagnosed disorder of amino or organic acid metabolism

Ages: 2 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: Children with PKU and age- and sex-matched non-PKU comparison subjects.
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Amino acid levels in blood | day 1
  Measuring amino acid levels in blood [μmol/L]
Nutrient Intake | day 1 - day 3
  Measured by three-day diet diary. Nutrients in [mg/day]

CONTACTS AND LOCATIONS:
Overall Officials: Dr. P. Verloo, Principal Investigator — UZ Gent, Belgium
Locations (2):
- Dr. P. Verloo, Ghent, Belgium
- Birmingham Children's Hospital, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No